CLINICAL TRIAL: NCT06274892
Title: Remote Monitoring of Patient Reported Outcomes to Improve the Efficacy of the Acute Phase Radiotherapy Review Process
Acronym: PROMOTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-5818
Record Dates: First submitted 2023-10-25; First posted 2024-02-23 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Breast Cancer
Keywords: Radiation Therapy; Patient reported outcomes; Remote monitoring; Mobile phone application
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote monitoring PROs (Experimental): All participants allocated to the interventional arm will receive the RT technique, dose and fractionation according to institutional standards. Once per week, participants will use a mobile phone 'app' to enter mPROs, and indicate a need for review for any other reason. The treatment Radiation Therapists will triage the participant to either attend or skip that week's on-treatment review based on this information and established criteria. After RT completion, Advanced Practice Radiation Therapists (apRTs) will triage the participant to receive a virtual follow-up visit when necessary. Participants will be seen once by a Radiation Oncologist 4 to 12 weeks after last radiation treatment. The participants will also complete the following questionnaires: 1) Baseline (patient factors); 2) 'During treatment' (review quality); 3) 'Post acute phase' (satisfaction with care). Circle-of-care HCP will comment on the impact of the PROMOTE process on the quality of care for that participant.
  Interventions: Other: Remote monitoring PROs
- Standard of Care (No Intervention): All participants allocated to the standard of care arm will receive all RT treatment activities according to institutional standards. Participants will attend the weekly in-person review session with a Radiation Oncologist during treatment and will be seen once between 4 and 12 weeks after last RT treatment. Documentation of radiation-related toxicity will be performed by the radiation HCPs according to standard of care. Participants will be asked to complete the following study questionnaires: 1) Baseline evaluation (patient factors); 2) 'During treatment' evaluation (need/usefulness of review); 3) 'Post acute phase' evaluation (satisfaction with care).

INTERVENTIONS:
Other: Remote monitoring PROs — Attendance at RT review appointments triaged based on remotely monitored PROs
  Other Names: Zamplo mobile healthcare application
  Arms: Remote monitoring PROs

SUMMARY:
Radiation therapy (RT) is a key component in the treatment of breast and prostate cancer. However, patients may experience significant side effects. Patients can accurately self-report side effects from RT and these patient-reported outcomes (PROs) can direct communication between patient and healthcare provider (HCP), and facilitate joint decision making.

Patients state that using mobile phone applications (apps) to collect PROs (mPROs) is easily incorporated into their daily routines, allowing them to engage at a time and pace that suits them. When mPRO collection is combined with remote symptom monitoring by HCPs, these systems result in improvements in symptom control and quality of life.

Currently, patients receiving RT are seen by a Radiation Oncologist once per week during RT and once every few months after RT has finished. Recent evaluations indicate that patients and physicians consider the number of visits to be too frequent during RT, and too infrequent immediately after RT. This research will use weekly mPROs (remotely monitored by RT HCP) to determine if a patient needs (or wants) to be seen by a RT HCP during and/or immediately after RT.

Using mPROs to optimize RT patient assessment processes will ensure patients are seen if and when required. For a patient, this could result in reduced time and costs at the hospital. For the physician, resources could be re-allocated to improve access to RT services. Using mPROs after RT has the potential for earlier treatment of side effects, which has been linked to improved survival and quality of life.

DETAILED DESCRIPTION:
Rationale: Remote monitoring of mPROs provides a platform for near real-time monitoring and action, resulting in the systematic reporting of symptoms and the potential for earlier healthcare interventions to treat those symptoms. The use of mPRO monitoring has been linked to improved survival and quality of life in patients receiving chemotherapy. It is likely therefore, that similar benefits will be seen in RT, particularly in the period immediately after RT has finished.

In this study, the collection of mPROs will inform decision making when determining if a patient should be seen by a radiation oncologist. This will ensure patients in need of care are seen in a timely manner, if and when required. For a patient and caregiver, reduced time at the hospital leads to reduced opportunity costs (e.g. time) and out-of-pocket fees (e.g. parking). For the physician, the work time and clinic space gained from not seeing 'well' patients can be re-allocated to seeing 'unwell' patients or seeing new patient consultations to improve access to RT services. Hence, remotely monitoring mPROs to shape RT supportive care processes may reduce costs for patients and improve efficiency for physicians without a detrimental impact on quality of care.

To date, no research has evaluated the use of remote monitored mPROs to triage RT patients' supportive care, based on patient assessments of need. It is hypothesized that the use of remote mPRO monitoring will reduce the number of in-person review visits during RT and/or improve patient care immediately after RT.

Objectives: Primary) To determine if remote mPRO monitoring influences the proportion of review visits necessary during and up to 12 weeks after RT. Secondary) To determine the patient and treatment factors that influence the number and pattern of radiation HCP assessments needed during and up to 12 weeks after RT; to quantify the impact of mPRO remote monitoring on the frequency of adverse events and the use of unscheduled acute care services.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast or prostate cancer
* About to receive a course of radical or adjuvant radiation therapy as an outpatient at Princess Margaret Cancer Centre
* Able to enter PRO responses into the mobile app in English or French

Exclusion Criteria:

* Significant comorbidities that would render the patient not suitable for remote monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Remote monitoring efficiency | At the end of radiation (average 5 weeks), and 12 weeks after completion of radiation
  Proportion of review visits attended during RT, and up to 12 weeks after RT. Number of review visits attended (from weekly participant questionnaire) as a percentage of the total possible review visits.
  Values will range from 0% to 100%. Low percentage indicates desirable outcome.

SECONDARY OUTCOMES:
Remote monitoring efficacy | At the end of radiation (average 5 weeks), and 12 weeks after completion of radiation
  Frequency of Grade 2 or above toxicity (PRO-CTCAE v1) (from mPRO entries)
Remote monitoring value | At the end of radiation (average 5 weeks)
  Patient assessment of review 'value' (from weekly participant questionnaire) for each review visit attended.
  Question asked "Was the review session a valuable use of your time?". Response options: 4 point Likert scale "Not at all, A little bit, Quite a bit, Very much".
  Values will range from 0 to 3. High score indicates desirable outcome.
Remote monitoring comprehensiveness | At the end of radiation (average 5 weeks), and 12 weeks after completion of radiation
  Number of times unscheduled acute care services were used (from questionnaire)
Influencing factors (patient) | At the end of radiation (average 5 weeks)
  Sociodemographic factors (from questionnaire) associated with the proportion of review visits attended
Influencing factors (disease) | At the end of radiation (average 5 weeks)
  Disease factors (from chart review) associated with the proportion of review visits attended
Influencing factors (treatment) | At the end of radiation (average 5 weeks)
  Treatment factors (from chart review) associated with the proportion of review visits attended
Influencing factors (toxicity) | 12 weeks after completion of radiation
  Frequency of Grade 2 or above toxicity (PRO-CTCAE v1) 'during RT' associated with the proportion of 'after RT' review visits

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan